CLINICAL TRIAL: NCT05983471
Title: A Randomized, Double-blind, Placebo-controlled, Cross-over Trial to Evaluate the Efficacy and Safety of ME-015 (Suplatast Tosilate) in Cough Related to Idiopathic Pulmonary Fibrosis
Brief Title: Efficacy and Safety of ME-015 (Suplatast Tosilate) in Cough Related to Idiopathic Pulmonary Fibrosis (COSMIC-IPF)
Acronym: COSMIC-IPF
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Melius Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COSMIC-IPF; SYNCD-070-22 (Other: Syngene International)
Record Dates: First submitted 2023-07-24; First posted 2023-08-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Idiopathic Pulmonary Fibrosis; Cough; IPF; Fibrotic Lung Disease; Chronic Cough; Coughing
Keywords: IPF-cough; IPF cough; Idiopathic Pulmonary Fibrosis; Chronic cough; Suplatast; Melius; Refractory cough; IPF; Fibrotic cough; Melius Pharma; RCT; Sequential; Cough frequency; Cough severity; India; fibrosis; Oral; New Chemical Entity; Small molecule; Nowak; Kornfeld; Sweden
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Cough; Chronic Cough; Fibrosis | interventions — MO 113; suplatast tosilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Interactive web response system (IWRS)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm 1 (Experimental): 2 weeks of blinded active treatment, followed by 2 weeks of blinded placebo treatment (wash-out), followed by 2 weeks of blinded placebo treatment, followed by 1 week of follow-up with neither active nor placebo treatment
  Interventions: Drug: ME-015 (Suplatast Tosilate); Other: Identical placebo
- Treatment Arm 2 (Experimental): 2 weeks of blinded placebo treatment, followed by 2 weeks of blinded placebo treatment (wash-out), followed by 2 weeks of blinded active treatment, followed by 1 week of follow-up with neither active nor placebo treatment
  Interventions: Drug: ME-015 (Suplatast Tosilate); Other: Identical placebo

INTERVENTIONS:
Drug: ME-015 (Suplatast Tosilate) — Oral capsule form, 200 mg t.i.d. (total 600 mg per 24 hours)
  Other Names: Suplatast; Suplatast Tosilate
Other: Identical placebo — Without active component

SUMMARY:
Orally administered ME-015 (Suplatast Tosilate) has been available on the market as a prescription drug for allergy-related conditions in Japan since 1995 with a good safety and tolerability profile.

There is preclinical and exploratory clinical evidence suggesting that ME-015 may be effective in treating cough caused by idiopathic pulmonary fibrosis (IPF cough).

80% of patients with idiopathic pulmonary fibrosis (IPF) are affected by a devastating dry cough that is often not responsive to standard cough treatments and causes significant psychological and physiological suffering as well as reduced quality of life. As of November 2024, there is no approved treatment for IPF cough. There is an enormous unmet clinical need for an effective, safe and well-tolerated oral treatment; particularly as approved antifibrotic treatments (pirfenidone and nintedanib) have not been shown to reduce cough in controlled clinical trials.

The COSMIC-IPF Phase 2a trial is the first clinical trial assessing ME-015 (an NCE outside of Japan) for the treatment of IPF cough and aims to generate clinical proof-of-concept results regarding the safety and efficacy of ME-015 in this condition.

DETAILED DESCRIPTION:
This quadruple blinded, cross-over, placebo-controlled clinical trial will randomize patients with stable idiopathic pulmonary fibrosis (IPF) and cough related to IPF (IPF cough) in a 1:1 fashion to one of two treatment sequences: active treatment followed by placebo, or placebo followed by active treatment. Each 14-day active/placebo treatment phase is preceded by a wash out period. The treatment sequences are followed by an observational 7-day follow-up period without medication. All subjects in the trial receive standard-of-care antifibrotic treatment for IPF. There is a single-blinded placebo run-in period before randomization to create a stable baseline and adjust for the anticipated placebo effect at study entry.

Treatment assignment is blinded to patients, investigators, site personnel, data analysts and Sponsor. The active treatment is ME-015 (Suplatast Tosilate) 200 mg t.i.d. (three times per day) administered as oral capsules. The placebo treatment consists of identical capsules without the active component.

The primary efficacy endpoint is the effect on awake time cough frequency measured objectively with the VitaloJak device over a 24-hour period. VitaloJak recordings are analysed using a blinded, independent, central review and validation process.

The study is conducted as a single-country, multi-centre clinical trial in India with Melius Pharma AB as the Sponsor. External central adjudication of HRCT images by a UK-based KOL ensures guideline-based diagnoses of IPF. Treatment needs to follow international guideline-based standard of care for IPF, and all Indian sites have been chosen to reflect a similar standard of care as practiced in Europe and the U.S. Only literate patients are enrolled into the trial and all patient-facing material is made available in English and all common local languages.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of IPF according to 2018 ATS/ERS/JRS/ALAT guidelines, confirmed by high-resolution computed tomography (HRCT) chest scan taken < 2 years ago
2. Age ≥ 18 years
3. Cough attributed to IPF unresponsive to standard anti-tussive treatment and present for > 8 weeks
4. Arithmetic mean of ≥ 10 coughs/hour during waking hours
5. Ability to read, comprehend, and complete the ICF and all questionnaires in the study without help
6. Cough severity score of ≥ 40 mm on a 0-to-100 mm Visual Analogue Scale (VAS)
7. Willing and able to comply with the protocol
8. Life expectancy > 6 months
9. Stable medical condition: stable treatment for > 12 weeks and absence of acute exacerbations for > 4 weeks
10. FVC ≥ 40% predicted
11. FEV1 / FVC ≥ 65%
12. Women of childbearing potential must agree to use a highly effective method of contraception
13. Male partner must agree to use a condom during the study, unless they had a vasectomy > 6 months prior to first study drug administration

Exclusion Criteria:

1. Likely need for lung transplantation in next 12 months
2. Permanent long-term oxygen therapy
3. Use of high-dose corticosteroids or cytotoxic medications
4. History of unstable or deteriorating cardiac or pulmonary disease in the preceding 6 months
5. Current smoking, vaping, or tobacco chewing
6. Treatment with an ACE inhibitor or sitagliptin
7. Any antitussive treatment, including opioid-based and OTC, for treatment of cough within 4 weeks of Screening or at any point during the study
8. BMI < 18 kg/m2 or ≥ 40 kg/m2
9. Suspected acute infection, including COVID-19 or influenza or any upper respiratory tract infection
10. History of malignancy within the last 2 years
11. History of drug/ alcohol dependency/ abuse within the last 2 years
12. Condition that could affect drug absorption
13. Recent history of stroke or TIA
14. Resting blood pressure > 160/90 mmHg
15. Pregnant/lactating women
16. Investigational drug or biologic within the last 2 months
17. Blood donation within the last 56 days or plasma donation within the last 7 days
18. Severe medical/ psychiatric condition posing risk to trial participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Wake time cough frequency during 24 hours | Change from Baseline to Day 14 in the respective treatment period
  Measured objectively over a 24-hour period with the cough recording device VitaloJak and processed using centralized, blinded, QC'd analysis

SECONDARY OUTCOMES:
Cough severity in the last 24 hours | Change from Baseline to Day 14 in the respective treatment period
  Visual Analogue Scale (VAS) ranging from 0 - 100 mm where higher values indicate more severe cough
Cough-related quality of life in the last 24 hours | Change from Baseline to Day 14 in the respective treatment period
  Leicester Cough Questionnaire (LCQ) total score ranging from 3 - 23 where lower values indicate greater impairment of health status due to cough
Overall patient-reported health status | Change from Baseline to Day 14 in the respective treatment period
  Global Rating of Change Scale of cough severity (range -7 to +7) and cough frequency (range -7 to +7) where 0 indicates no change, higher values above 0 indicate larger improvement, and lower values below 0 indicate increased declined
Safety: Treatment-Emergent Adverse Events | From enrolment into the trial until end of follow-up, circa 50-60 days per subject
  Incidence of treatment-emergent adverse events (TEAE)
Safety: Adverse Events and Serious Adverse Events | From enrolment into the trial until end of follow-up, circa 50-60 days per subject
  Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Safety: Vital Signs - blood pressure | From enrolment into the trial until end of follow-up, circa 50-60 days per subject
  Resting blood pressure (mmHg), assessed weekly
Safety: Vital Signs - heart rate | From enrolment into the trial until end of follow-up, circa 50-60 days per subject
  Heart rate (bpm) - assessed weekly during the trial
Safety: Vital Signs - body temperature | From enrolment into the trial until end of follow-up, circa 50-60 days per subject
  Body temperature (degrees Celsius) - assessed weekly during the trial
Safety: Clinical Laboratory Results | From enrolment into the trial until end of follow-up, circa 50-60 days per subject
  Clinical laboratory results (chemistry, hematology, urine dipstick) analysed by a central laboratory

OTHER OUTCOMES:
Exploratory Endpoint: 24-hour Cough Frequency | Change from Baseline to Day 14 in the respective treatment period
  24-hr cough frequency recording with the VitaloJak device and analysed using central, blinded review and QC
Exploratory Endpoint: Sleep-time Cough Frequency | Change from Baseline to Day 14 in the respective treatment period
  Sleep-time cough frequency based on 24-hour recording with the VitaloJak device and analysed using central, blinded review and QC
Exploratory Endpoint: Patient-Reported Breathlessness | Change from Baseline to Day 14 in the respective treatment period
  Patient-reported outcome breathlessness assessed using the 12-item Dyspnoea-12 Questionnaire
Exploratory Endpoint: Patient-reported Cough Hypersensitivity | Change from Baseline to Day 14 in the respective treatment period
  Patient-reported outcome assessed using the Cough Hypersensitivity Questionnaire (CHQ)
Exploratory Endpoint: Eosinophilia | Change from Baseline to Day 14 in the respective treatment period
  Eosinophil count (total and % of white blood cells in peripheral blood) measured using a central laboratory
Exploratory Endpoint: Pulmonary Function | Change from Baseline to Day 14 in the respective treatment period
  Pulmonary function assessed using local spirometry assessments; specifically forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), and ratio of FEV1/FVC
Exploratory Endpoint: ME-015 Concentration in Blood | Change from Baseline to Day 14 in the respective treatment period
  Concentration of ME-015 and its major metabolie M-1 is peripheral blood samples taken once at each visit alongside safety lab samples

CONTACTS AND LOCATIONS:
Locations (6):
- India (6):
  - Aditya Multi Specialty Hospital, Guntur, Andhra Pradesh
  - KLE's Dr Prabhakar Kore Hospital & Medical Research Centre, Belagavi, Karnataka
  - ACE Hospital and Research Centre, Pune, Maharashtra
  - Hindusthan Hospital, Coimbatore, Tamil Nadu
  - GSVM Medical College, Murari Lal Chest Hospital, Kanpur, Uttar Pradesh
  - Health Point Hospital, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — https://www.meliuspharma.com/